CLINICAL TRIAL: NCT02938845
Title: Factors Related to Patients' Anxiety Before and After Hysterectomy
Brief Title: Does Minimally Invasive Surgery Reduce Anxiety?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Eser, medical doctor, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 025
Record Dates: First submitted 2016-10-12; First posted 2016-10-19 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- total laparoscopic hysterectomy(TLH) (Experimental): Each patient's anxiety was measured using Spielberger's State-Trait Anxiety Inventory immediately before, immediately after the operation.
  Interventions: Behavioral: Spielberger's State-Trait Anxiety Inventory(STAI ); Procedure: total laparoscopic hysterectomy(TLH)
- total abdominal hysterectomy(TAH) (Experimental): Each patient's anxiety was measured using Spielberger's State-Trait Anxiety Inventory immediately before, immediately after the operation.
  Interventions: Behavioral: Spielberger's State-Trait Anxiety Inventory(STAI ); Procedure: total abdominal hysterectomy(TAH)

INTERVENTIONS:
Behavioral: Spielberger's State-Trait Anxiety Inventory(STAI ) — State anxiety (STAI-S) refers to a temporary emotional state related to a specific situation, whereas trait anxiety (STAI-T) represents anxiety as a relatively stable personality character. Each scale has values ranging from 20 to 80, with higher scores representing more severe anxiety. The STAI has no established categories, but a cutoff score of 40 has been used to identify patients with high/very high anxiety. The validity and reliability of the Turkish versions of these instruments have been validated.
Procedure: total laparoscopic hysterectomy(TLH)
  Arms: total laparoscopic hysterectomy(TLH)
Procedure: total abdominal hysterectomy(TAH)
  Arms: total abdominal hysterectomy(TAH)

SUMMARY:
The purpose of this study was to identify factors that may contribute to anxiety of patients undergoing total abdominal hysterectomy(TAH) or total laparoscopic hysterectomy(TLH) before and after the operation. Thus, we aimed to learn whether anxiety levels change according to the type of hysterectomy.

DETAILED DESCRIPTION:
Hysterectomy is the most common gynecological procedure worldwide. . There has been a increasing interest towards to more minimally invasive procedures in the past decade. Hysterectomy operation anxiety is a complex phenomenon affected by various parameters. Patients' anxiety may be affected by their age, gender, educational status,type of operation and personality. Each patient's anxiety was measured using Spielberger's State-Trait Anxiety Inventory immediately before, immediately after the operation.

ELIGIBILITY:
Inclusion Criteria:

undergone hysterectomies for benign reasons.

Exclusion Criteria:

malignancy, additional operation beside hysterectomy( such as salpingo-oophorectomy), history of two or more previous caesarean sections, history of previous abdominal surgery, autoimmune disease, coagulation disorders, with known systemic or psychiatric disease, those receiving any regular sedative medication at the time of the procedure

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
STAI-S's Inventory | change from immediately before operation to immediately after the operation.
STAI-T's Inventory | change from immediately before operation to immediately after the operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Woman and Child Diseases Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Lopez-Jornet P, Camacho-Alonso F, Sanchez-Siles M. Assessment of general pre and postoperative anxiety in patients undergoing tooth extraction: a prospective study. Br J Oral Maxillofac Surg. 2014 Jan;52(1):18-23. doi: 10.1016/j.bjoms.2013.01.004. Epub 2013 Jan 26. PMID 23357053
- [Result] Muglali M, Komerik N. Factors related to patients' anxiety before and after oral surgery. J Oral Maxillofac Surg. 2008 May;66(5):870-7. doi: 10.1016/j.joms.2007.06.662. PMID 18423273
- [Result] Flory N, Bissonnette F, Binik YM. Psychosocial effects of hysterectomy: literature review. J Psychosom Res. 2005 Sep;59(3):117-29. doi: 10.1016/j.jpsychores.2005.05.009. PMID 16198184